CLINICAL TRIAL: NCT01454895
Title: Test of a Web-based Intervention to Promote Hearing Protector Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marjorie McCullagh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Marjorie McCullagh, Associate Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 00027046
Record Dates: First submitted 2011-10-14; First posted 2011-10-19 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Noise-induced Hearing Loss
Keywords: noise-induced hearing loss; prevention; farmers
MeSH Terms: conditions — Hearing Loss, Noise-Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Interactive Web-based Info (IWI) & HPDs (Experimental): Subjects will receive interactive Web-based information regarding farm noise exposures, risks to hearing, and strategies for protecting hearing, as well as a mailed sample of various types of hearing protection devices.
  Interventions: Behavioral: Sampler of hearing protection devices; Behavioral: Interactive Web-based information
- Interactive Web-based Information (IWI) (Experimental): This intervention includes a number of features/techniques designed to promote behavior change. Messages focus on farmer-friendly techniques for adopting use of HPDs. The factors found to be significant predictors of HPD use (Barriers to Use and Situational Factors Influencing HPD Use) are particularly relevant to farmers' learning needs, and are especially emphasized in this model-based intervention to increase hearing protector use among farmers. Participants will select the sequence of features they visit, as well as the time spent in each feature and number of visits to the site. Their patterns of use will be tracked by the enrollment and data collection systems and used in analysis.
  Interventions: Behavioral: Interactive Web-based information
- Static Web information (SWI) & HPDs (Experimental): Subjects will receive static Web-based information regarding farm noise exposures, risks to hearing, and strategies for protecting hearing, as well as a mailed sample of various types of hearing protection devices.
  Interventions: Behavioral: Sampler of hearing protection devices; Behavioral: Static Web-based information
- Static Web information only (Active Comparator): Subjects will receive interactive Web-based information regarding farm noise exposures, risks to hearing, and strategies for protecting hearing.
  Interventions: Behavioral: Static Web-based information
- Hearing protection Devices only (Experimental): Subjects will receive a mailed sample of various types of hearing protection devices.
  Interventions: Behavioral: Sampler of hearing protection devices
- Interactive Web-based information only (Other): used for cases enrolling after achievement of study enrollment goal
  Interventions: Behavioral: Interactive Web-based information

INTERVENTIONS:
Behavioral: Sampler of hearing protection devices — In a pilot study, hearing protection devices were mailed to farmers, resulting in a significant increase in use. These results suggested that overall, HPDs were acceptable to farmers, and that access to HPDs may be an important contributor to frequency of use. The study will build on this earlier work by providing an assortment of hearing protection devices to a sub-sample of each group of farmers receiving the Interactive and Static Web Interventions. The assortment includes the most commonly used types of devices (i.e., muffs, foam plugs, pre-molded plugs, and semi-aurals). The sampler is delivered, together with manufacturers' standard written instructions for use, via mail at the designated time according study design.
  Other Names: HPDs
  Arms: Hearing protection Devices only; Interactive Web-based Info (IWI) & HPDs; Static Web information (SWI) & HPDs
Behavioral: Static Web-based information — The standard information promoting HPD use delivered via Internet will be based on an informational brochure previously developed for use by farmers (i.e., Have You Heard? and They're Your Ears Protect Them). These brochures, including color graphics and text, are available on the Internet (as PDF files). Although they have been printed and distributed by NIOSH, most farmers will not have been exposed to copies. There are important differences between the SWI and IWI interventions, including interactivity, animation, explication of farmer-generated tips and techniques for addressing common barriers to hearing protector use, use of color, audio, and video, hotlinks, and farmer testimonials.
  Other Names: SWI
  Arms: Static Web information (SWI) & HPDs; Static Web information only
Behavioral: Interactive Web-based information — This intervention includes a number of features/techniques designed to promote behavior change. Messages focus on farmer-friendly techniques for adopting use of HPDs. The factors found to be significant predictors of HPD use (Barriers to Use and Situational Factors Influencing HPD Use) are particularly relevant to farmers' learning needs, and are especially emphasized in this model-based intervention to increase hearing protector use among farmers. Participants will select the sequence of features they visit, as well as the time spent in each feature and number of visits to the site. Their patterns of use will be tracked by the enrollment and data collection systems and used in analysis.
  Other Names: IWI
  Arms: Interactive Web-based Info (IWI) & HPDs; Interactive Web-based Information (IWI); Interactive Web-based information only

SUMMARY:
The purpose of this project is to compare the effectiveness of several approaches to influencing hearing protector use. The goals of this study are to further develop an intervention to promote farmers' use of hearing protectors, and compare the effectiveness of the developed intervention with two alternative approaches to influencing hearing protector use behavior, delivered in various combinations. This study will determine if significant change in hearing protection use can be achieved in a one-shot web-based or protector-supply intervention. Results will determine the need for future program modifications, e.g., inclusion of booster(s).

DETAILED DESCRIPTION:
OBJECTIVE: To further develop and test an intervention to promote farmers' use of hearing protection devices (HPDs).

SPECIFIC AIMS: The specific aim of this study is to contrast the effects of three alternative NIHL-prevention intervention strategies, delivered in various combinations on HPD use and use-related attitudes/beliefs. Specifically, the three approaches include: a) an interactive, predictors-based intervention delivered via the Internet ("Interactive Web," IWI); b) a static informational Web site designed to increase farmers' use of HPDs ("Static Web," SWI); and c) sampler of HPDs, e.g., ear muffs, plugs ("HPD Intervention," HPD I).

HYPOTHESIS 1: Participants receiving interactive Web interventions (IWI) will have higher hearing protector device (HPD) use and more favorable use-related attitudes/beliefs than participants not receiving interactive web interventions (IWI); HYPOTHESIS 2: Participants receiving the HPD intervention (HPDI)will have higher HPD use and more positive use-related attitudes/beliefs than participants not receiving the HPD intervention (HPDI). HYPOTHESIS 3: Participants visiting the Web site more frequently will have higher HPD use than those visiting less frequently. HYPOTHESIS 4. There will be no interaction between intervention delivery mode (interactive vs. static) and HPDI.

BACKGROUND: Farmers are among the most noise-exposed group of workers, and experience rates of noise-induced hearing loss (NIHL) of up to 72% compared to workers in other industries (x%). NIHL is associated with negative impact on quality of life, including difficulty in communication, risk of not hearing warning sounds, and tinnitus. Although use of hearing protection devices (HPDs) would protect them from NIHL, use among farmers is low. An earlier study identified predictors of use of HPDs as barriers, situational factors and gender, and accounted for 74% of the variance in use. These results also showed that a small proportion of farmers have successfully developed a variety of methods to overcome barriers and situational factors that interfere with HPD use. This project builds on the earlier work by applying these findings to develop a targeted intervention that also incorporates videotaped messages from the actual farmers who were frequent users of HPDs.

METHODS: The interventions, based on the Pender Health Promotion Model, will consist of Internet-based brief interactive motivational packages regarding adopting HPD use behaviors. Outcome measures will include self-reported frequency of HPD use, measured at 6 and 12 months post-intervention. The study will involve six experimental conditions. In the first condition, farmers will receive the interactive Web intervention (IWI) and an assortment of hearing protection devices (HPDs); in the second condition, farmers will receive the interactive Web intervention (IWI) only; in the third condition, farmers will receive the static Web intervention (SWI) and HPDs; in the fourth condition, farmers will receive the static Web intervention (SWI) only; in the fifth condition, farmers will receive the assortment of HPDs only. A sixth condition will deliver the interactive Web intervention only to farmers who enroll after the target of 709 enrollees, and will receive this service as a courtesy to the American Farm Bureau and its affiliates, but cases 710 and beyond will not receive incentives.

ELIGIBILITY:
Inclusion Criteria:

* farm operators who are active in production at least half-time,
* speak English
* at least 18 years of age
* have Internet access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2011-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Hearing protector device (HPD) use | 12 months

SECONDARY OUTCOMES:
hearing protector use-related attitudes/beliefs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie C. McCullagh, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] McCullagh MC, Banerjee T, Cohen MA, Yang JJ. Effects of interventions on use of hearing protectors among farm operators: A randomized controlled trial. Int J Audiol. 2016;55 Suppl 1(0):S3-12. doi: 10.3109/14992027.2015.1122239. Epub 2016 Jan 14. PMID 26766172
- [Derived] McCullagh MC, Ronis DL. Protocol of a randomized controlled trial of hearing protection interventions for farm operators. BMC Public Health. 2015 Apr 18;15:399. doi: 10.1186/s12889-015-1743-0. PMID 25927191